CLINICAL TRIAL: NCT02662140
Title: Mobile Health Solutions for Behavioral Skill Implementation Through Homework
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-01854
Record Dates: First submitted 2016-01-08; First posted 2016-01-25 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Oppositional Defiant; Conduct Disorder
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile Health Application Group (Experimental): emobile health application will enhance the existing evidence informed curriculum of a Multiple Family Group model (called 4 Rs and 2 Ss for Strengthening Families Model) for families with children who have disruptive behavior disorders. This mobile application consists of two primary components that will support engagement and integration of the model's core concepts in family life. The first component focuses on delivering HW via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process of HW. The second component focuses on targeting factors putatively related to poor HW implementation within the "Do" process.
  Interventions: Behavioral: Mobile Health Applictaion

INTERVENTIONS:
Behavioral: Mobile Health Applictaion — Component 1: Delivering homework via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process of HW.
  Component 2: Focuses on targeting factors putative related to poor HW implementation within the "Do" process

SUMMARY:
The primary purpose of this study is to develop a mobile health (mHealth) application that will both advance theory in and clinical practice of homework (HW) implementation. The mobile health application will enhance the existing evidence informed curriculum of a Multiple Family Group model (called 4 Rs and 2 Ss for Strengthening Families Model) for families with children who have disruptive behavior disorders. This mobile application consists of two primary components that will support engagement and integration of the model's core concepts in family life. The first component focuses on delivering homework via a highly engaging, multiplayer, interactive, cooperative, and skill-building game platform aimed at improving the "Design" and "Do" process of homework.The second component focuses on targeting factors putatively related to poor HW implementation within the "Do" process.

ELIGIBILITY:
Inclusion Criteria:

* youth between the ages of 7 to 11 years and an accompanying adult primary caregiver available to participate in the research and intervention activities
* English speaking youth and adult caregiver and
* the child should meet criteria for a primary diagnosis of Oppositional Defiant or Conduct Disorder.

Exclusion Criteria:

* a significant cognitive impairment or emergent psychiatric needs of the caregiver or child that interferes with understanding of program content or informed consent process or requires a higher level of care.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Demographics | 4 Months
  Demographics Interview
Measure of Disruptive Behavior Disorder (DBD) Symptoms using DBD Rating Scale | 4 Months
Measure of Child's Impairment using the Impairment Rating Scale | 4 Months
Change in quantity and quality of homework measured using the Homework Rating Scale -II | 4 Months
Change in Homework Adherence and Competence Scales | 4 Months
Change in Attendance to sessions | 4 Months
Change in Consumer Satisfaction and Feedback Measured by Weekly Interviews | 4 Months
Change in behavior measured by the IOWA Conners Oppositional/Defiant Scale | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mary McKay, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States